CLINICAL TRIAL: NCT05902364
Title: Systane® Ultra Preservative Free Lubricant Eye Drops
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DEU894-I001
Record Dates: First submitted 2023-06-02; First posted 2023-06-15 (Actual); Results first posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 - Dry Eye Symptoms (Experimental): 1-2 drops of Systane Ultra PF lubricant eye drops in each eye four times a day for 30 days
  Interventions: Other: Systane Ultra PF lubricant eye drops
- Group 2 - CL-Related Dryness Discomfort (Experimental): 1-2 drops of Systane Ultra PF lubricant eye drops in each eye four times a day for 30 days
  Interventions: Other: Systane Ultra PF lubricant eye drops

INTERVENTIONS:
Other: Systane Ultra PF lubricant eye drops — Commercially available preservative free eye drops
  Other Names: Systane Ultra Preservative-Free

SUMMARY:
The purpose of this post-market clinical follow-up (PMCF) study is to assess the performance and safety of Systane Ultra Preservative-Free (PF) in subjects experiencing dry eye symptoms (Group 1) and contact lens (CL) wearers experiencing discomfort due to CL-related dryness (Group 2). Statistical analyses will be presented by group. This study will be conducted in Canada, Australia, and New Zealand.

DETAILED DESCRIPTION:
Subjects will participate in the study for approximately 30 days, with a phone call scheduled on Day 15 ± 2 (Visit 2) and a follow-up visit scheduled on Day 30 ± 2 (Visit 3). Subjects will be asked to complete patient questionnaires on Day 1 and at Visit 3 (Impact of Dry Eye on Everyday Life - Symptom Bother [IDEEL-SB] or Contact Lens Dry Eye Questionnaire [CLDEQ-8] and Comfortable Wear Time questions).

ELIGIBILITY:
Inclusion Criteria:

* Subject must be able to understand and sign an informed consent form.
* Subject with mild to moderate dry eye.
* Subject with contact lens-related dry eye symptoms.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Has suffered any ocular injury to either eye in the past 3 months prior to screening.
* Has undergone any other ocular surgery (including intraocular surgery) within the past 6 months or has any ocular surgery planned during the study.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2023-10-28 (Actual); Primary Completion 2024-08-14 (Actual); Study Completion 2024-08-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Lead, Vision Care, Study Director — Alcon Research, LLC
Locations (4):
- Canada (2):
  - Integra Eye Care, Burnaby, British Columbia
  - University of Waterloo School of Optometry, Waterloo, Ontario
- New Zealand (2):
  - University of Auckland, Grafton, Auckland
  - Rose Optometry, Frankton, Otago

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 69 subjects enrolled in the study (signed an informed consent), 1 subject was determined to be ineligible and was exited from the study prior to treatment. This reporting group includes all eligible subjects.
Period: Overall Study
Arm/Group | Group 1 - Dry Eye Symptoms | Group 2 - CL-Related Dryness Discomfort
Started | 34 | 34
Completed | 33 | 34
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set: All subjects exposed to at least one dose of Systane Ultra PF
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 - Dry Eye Symptoms | Group 2 - CL-Related Dryness Discomfort | Total
Number analyzed (Participants) | 34 | 34 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.9 (17.15) | 35.2 (11.05) | 38.6 (14.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 29 | 57
  Male | 6 | 5 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 10 | 16 | 26
  Black or African American | 0 | 0 | 0
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0
  White | 14 | 8 | 22
  Multi-racial | 0 | 0 | 0
  Other | 2 | 3 | 5
  Unknown | 8 | 6 | 14
Region of Enrollment [Number; unit: participants]
  Canada | 24 | 15 | 39
  New Zealand | 10 | 19 | 29

OUTCOME MEASURES:

1. Primary Outcome: Mean Overall IDEEL SB Score - Group 1
Description: The Impact of Dry Eye on Everyday Life Symptom Bother (IDEEL SB) module is a 20-item, patient-reported outcome questionnaire that assesses the subject's symptoms of dry eye. For each item, the subject selected a single response for both eyes, where 0 = "None of the time" (Q1) or "I did not have this symptom/Not Applicable" (Q2-20) to 4 = "All of the time" (Q1) or "Very Much" (Q2-20). The overall score was calculated as the mean value of the non-missing item scores (Q1-20) multiplied by 25 and ranged from 0 (minimum) to 100 (maximum). Baseline was defined as the last non-missing value prior to the start date of the study treatment. For subjects who were not exposed, Baseline was defined as the value from Visit 1 (Screening). Higher scores indicate greater symptom bother. No statistical hypothesis was pre-specified for this endpoint. This endpoint was pre-specified for Group 1
Time Frame: Baseline (Day 1), Day 30
Population: Full Analysis Set with data at visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 - Dry Eye Symptoms
Number analyzed (Participants) | 33
score on a scale
  Day 1 | 45.53 (11.784)
  Day 30 | 31.23 (10.854)

2. Primary Outcome: Mean Overall CLDEQ-8 Score - Group 2
Description: The Contact Lens Dry Eye Questionnaire-8 (CLDEQ-8) is an 8-item, patient-reported outcome questionnaire that evaluates the severity of dry eye symptoms in soft contact lens wearers within the past 2 weeks. For each item, the subject selected a single response for both eyes using a 0-4, 0-5, or 1-6 Likert scale. The overall score was calculated as the sum of the numerical responses for each of the 8 items and ranged from 1 (minimum) to 37 (maximum). A lower CLDEQ-8 score indicates less frequent or less intense symptoms. Baseline was defined as the last non-missing value prior to the start date of the study treatment. For subjects who were not exposed, Baseline was defined as the value from Visit 1 (Screening). No statistical hypothesis is pre-specified for this endpoint. This endpoint was prespecified for Group 2 only.
Time Frame: Baseline (Day 1), Day 30
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 2 - CL-Related Dryness Discomfort
Number analyzed (Participants) | 34
score on a scale
  Day 1 | 19.4 (5.84)
  Day 30 | 10.3 (4.64)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from time of consent until study exit, approximately one month. AEs were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator. "At Risk" population for ocular AEs is reported in units of eyes; all other populations are reported in units of subjects. This analysis population includes all subjects/eyes exposed to any study lenses, as treated.
Description: All participants were monitored for serious and other ocular and nonocular AEs. All-Cause Mortality was not monitored for the ocular arms. However, the nonocular AE arms were not considered at risk for ocular adverse event terms as the arms are reporting nonocular-specific AEs. Similarly, the ocular AE arms were not considered at risk for nonocular adverse event terms as the arms are reporting ocular-specific AEs.
Groups:
- Group 1 - Ocular Adverse Events; Group 1 - Nonocular Adverse Events; Group 2 - Ocular Adverse Events; Group 2 - Nonocular Adverse Events: 1-2 drops of Systane Ultra PF lubricant eye drops in each eye four times a day for 30 days
Arm/Group | Group 1 - Ocular Adverse Events | Group 1 - Nonocular Adverse Events | Group 2 - Ocular Adverse Events | Group 2 - Nonocular Adverse Events
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/34 | 0/0 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/68 | 0/34 | 0/68 | 0/34
Other Adverse Events (participants affected / at risk) | 0/68 | 2/34 | 0/68 | 1/34
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Group 1 - Ocular Adverse Events (N=68) | Group 1 - Nonocular Adverse Events (N=34) | Group 2 - Ocular Adverse Events (N=68) | Group 2 - Nonocular Adverse Events (N=34)
Naspoharyngitis (Infections and infestations) | 0/0 | 2 | 0/0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2023-11-03): https://cdn.clinicaltrials.gov/large-docs/64/NCT05902364/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-29): https://cdn.clinicaltrials.gov/large-docs/64/NCT05902364/SAP_001.pdf